CLINICAL TRIAL: NCT06943469
Title: Synbiotics in Partially Hydrolysed Formula for Improved skiN Barrier Function in Infants at Risk for Allergy (SPHINX Study)
Brief Title: Effect of Partially Hydrolyzed Formula With Synbiotics on Skin Barrier Function
Acronym: SPHINX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2215INF
Record Dates: First submitted 2025-03-17; First posted 2025-04-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test formula (Experimental): Partially hydrolyzed formula with synbiotics
  Interventions: Other: Test formula
- Control formula (Active Comparator): Intact protein formula without synbiotics
  Interventions: Other: Control formula
- Reference arm (No Intervention): Breastfed arm (not applicable for France)

INTERVENTIONS:
Other: Test formula — Partially hydrolyzed formula with synbiotics
  Arms: Test formula
Other: Control formula — Intact protein formula without synbiotics
  Arms: Control formula

SUMMARY:
The main purpose of this study is to assess the efficacy of a partially hydrolyzed formula with synbiotics in halting one of the first steps of the allergic march (atopic dermatitis) in infants at risk of allergy. Other efficacy and safety parameters will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from at least one parent or legally acceptable representative (LAR), if applicable
2. Infant gestational age ≥ 37 completed weeks
3. Infant birth weight of ≥ 2.5 kg and ≤ 4.5 kg
4. Infant postnatal age ≤ 14 days (date of birth = day 0) at enrollment
5. Infant from singleton birth or infant from multiple births may if all birth siblings are enrolled.
6. At least one biological parent or sibling has (or had) a medically diagnosed history of allergy, based on response to a simple screening questionnaire
7. a. For the breastfed reference group only: infant is exclusively breastfed since birth with no intake of formula, and their parent(s) have the intention to continue exclusive breastfeeding until at least 4 months of age.

   or b. For the randomized formula-fed groups only: infant is exclusively or predominantly formula-fed in the 24 hours prior to enrollment, with formula feeding representing at least 75% of total daily feeds. The decision to introduce formula feeding was independently made by the parents before enrollment.
8. Parents/LAR must be able to provide evidence of parental authority and identity.
9. Infant's parent(s)/LAR must understand the informed consent form and other study documents and are willing and able to fulfill the requirements of the study protocol.

Exclusion Criteria:

1. Infectious, metabolic, congenital, genetic, gastrointestinal illness or any other condition (e.g., gastrointestinal surgery) that could impact oral feeding, growth or study outcomes.
2. Infants with special dietary needs other than standard infant formula (e.g., extensively hydrolyzed formula, amino acid formula, special formula for metabolic diseases) or requiring tube feeding.
3. Infant has already been diagnosed with allergy by a physician, including AD and/or cow's milk allergy.
4. Infant is currently participating or has previously participated in another clinical trial prior to enrollment.
5. Infant's parents or LARs have not reached legal age of majority (18 years).

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
TransEpidermal Water Loss (TEWL) at 3 months | At 3 months of age
  TransEpidermal water loss will be measured using a validated non-invasive technique.

SECONDARY OUTCOMES:
Cumulative incidence of Atopic Dermatitis | From enrollment to 12 months of age
  Cumulative incidence of AD is based on physician diagnosis using the United Kingdom Working Party (UKWP) diagnosis criteria.
TransEpidermal Water Loss | From enrollment to 12 months of age
  Epidermal water loss will be measured using a validated non-invasive technique.
Skin surface (stratum corneum) hydration | From enrollment to 12 months of age
  Skin hydration will be measured with a corneometer device.
Extent and severity of Atopic Dermatitis | From 3 months to 12 months of age
  SCORAD (SCORing for Atopic Dermatitis), scores range from 0 to 103, with higher scores indicating higher atopic dermatitis severity
Cumulative use of topical steroids and calcineurin inhibitors | From enrollment to 12 months of age
  Use of medication to treat AD and other symptoms will be collected via parent self-reported questionnaire.
Skin cytokines | From enrollment to 12 months of age
  Concentration of skin cytokines such as IL4 and IL5 using immunoassays
Skin natural moisturizing factors | From enrollment to 12 months of age
  Concentration of skin natural moisturizing factors such as Pyrrolidone carboxylic acid, using HPLC
Skin stratum corneum lipids | From enrollment to 12 months of age
  Concentration of skin stratum corneum lipids such as ceramides, cholesterol and triacylglycerol using mass spectrometry
Skin microbiome | From enrollment to 12 months of age
  Overall skin microbiome composition and diversity using next-generation sequencing
Skin metabolites | From enrollment to 12 months of age
  Levels of skin metabolites using targeted or untargeted approaches.
Immune proteomics | From enrollment to 6 months of age
  Levels of plasma proteins using mass cytometry or immunoassaysand immunoassays.
Immune blood cell immunophenotyping | From enrollment to 6 months of age
  Levels of immune cell populations using mass cytometry or immunoassays
Specific IgE antibodies | At 12 months of age
  Specific IgE antibodies will be measured using Phadiatop infant®.
Fecal microbiome | From enrollment to 12 months of age
  Overall fecal microbiota composition, diversity, different bacteria taxa and microbiota community types assessed using next generation sequencing (NGS) technology
Fecal metabolites | From enrollment to 12 months of age
  Levels of fecal metabolites using targeted or untargeted approaches.
Fecal biomarkers of inflammation and immunity | From enrollment to 12 months of age
  Levels of fecal markers of immune health and inflammation such as total secretory IgA (sIgA), calprotectin, and α-1-antitrypsin assessed by ELISA.
Physician-diagnosed allergic manifestations | From enrollment to 12 months of age
  Number of participants with Physician-diagnosed allergic manifestations.
Gastrointestinal tolerance | At enrollment and 4 months of age
  Infant Gastrointestinal Symptom Questionnaire (IGSQ), scores range from 13 to 65, with higher scores indicating higher gastrointestinal discomfort.
Weight | From enrollment to 12 months of age
  Weight (g and z-scores)
Height | From enrollment to 12 months of age
  Length (cm and z-scores)
Head circumference | From enrollment to 12 months of age
  Head circumference (cm and z-scores)
Safety assessment | From enrollment to 13 months of age
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (23):
- Belgium (3):
  - AZ Sint-Jan Brugge-Oostende AV - Campus Sint-Jan, Bruges
  - Universitair Ziekenhuis Brussel - Kinderziekenhuis, Brussels
  - Clinique Ste Elisabeth, Namur
- France (6):
  - CHU Amiens Picardie, Amiens
  - CHU de Caen, Caen
  - CHU de Grenoble Alpes, Grenoble
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Charles Nicolle, Rouen
  - CHRU de Tours, Tours
- Germany (5):
  - Charite-Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK), Berlin
  - Evangelisches Krankenhaus Düsseldorf - Frauenklinik, Düsseldorf
  - Klinik für Kinder- und Jugendmedizin, Universitätsklinikum Frankfurt, Frankfurt
  - Evangelisches Waldkrankenhaus Spandau, Spandau
  - Marien Hospital Wesel GmbH, Wesel
- Spain (9):
  - Hospital Teresa Herrera, A Coruña
  - HU Torrecárdenas, Almería
  - Hospital Quiron Salud Barcelona, Barcelona
  - Hospital Universitario Severo Ochoa, Madrid
  - Grupo Pediátrico Uncibay, Málaga
  - Instituto Hispalense de Pediatria (IHP), Seville
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari Sant Joan de Reus, Tarragona
  - HCU Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No